CLINICAL TRIAL: NCT00008892
Title: Anatomic MRI Brain Imaging of White Matter in Children
Brief Title: Brain Imaging in Children With AD/HD
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010064; 01-M-0064
Record Dates: First submitted 2001-01-18; First posted 2001-01-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-01-31

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Healthy
Keywords: Magnetic Resonance Imaging; Diffusion Tensor Imaging; Twin Study; Attention Deficit Hyperactivity Disorder; Normal Volunteers
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

SUMMARY:
The purpose of this study is to use brain imaging technology to study the connections between brain regions in children with attention deficit hyperactivity disorder (AD/HD), and comparing them to children without AD/HD.

This study will build upon previous brain imaging studies of healthy volunteers and children who have AD/HD. This study will use diffusion tensor magnetic resonance imaging (DT-MRI) to visualize and measure certain parts of the brains of identical twin pairs in which one twin has AD/HD, combined type.

Participants in this study will be screened with questionnaires and interviews, psychometric testing, and a physical examination. Participants' medical and educational records may be reviewed. Participants will undergo an MRI scan of the brain. Prior to the MRI, participants will have a training session in a simulated MRI scanner to learn how to lie still during MRI scanning. Participants may be asked to return for a follow-up scan in about 2 years.

DETAILED DESCRIPTION:
Attention-deficit/hyperactivity disorder (ADHD) is the most common childhood psychiatric disorder, present in between 3 to 10% of children in the United States (Wender et al 2001). It is thought to reflect subtle anomalies in the central nervous system and thus structural neuroimaging has been used extensively to delineate the neurobiology of the disorder. Magnetic resonance imaging has demonstrated structural anomalies in ADHD, affecting all the major lobes with particularly severe volume reductions in the cerebellum and relative preservation of the caudate nucleus (for a review see Durston 2003). In structural neuroimaging work, studies with monozygotic twins who are discordant for the disorder have proved a particularly powerful tool, with findings of a significantly smaller caudate nucleus in the affected twin compared to the unaffected, but genetically identical, twin (Castellanos et al 2003). We have previously reported an overall reduction in white matter volume in all four major brain lobes, with the deficit appearing to be fixed and non-progressive. However, recent advances in neuroimaging of white matter make feasible an examination of white matter characteristics, such as the degree of myelination and the coherence of white matter tracts. The proposed project builds on our anatomic magnetic resonance imaging (MRI) studies that have been performed with a 1.5-Tesla scanner in children who have Attention-Deficit/Hyperactivity Disorder (ADHD) and normal controls. We now propose to use diffusion tensor magnetic resonance imaging (DT-MRI) as conventional T(1)- and T(2)-weighted images at 3-Tesla to visualize and quantify white matter tracts in the brains of normal monozygotic (MZ) twins, MZ twins who are concordant for ADHD, and MZ twins who are discordant for ADHD. Ages will range from 6 to 21 years. Our principal focus will be on development and possible abnormalities of white matter tracts linking prefrontal-striatal-thalamic circuits in which we hypothesize disruption of these tracts in affected twins relative to their healthy co-twins. We will also explore the usefulness of this technique in delineating white matter in cerebellar circuits and characterize the normal development of white matter from ages 6 to 21 by using a single healthy twin per family.

ELIGIBILITY:
* INCLUSION CRITERIA:

PILOT SUBJECTS:

Subjects for pilot data collection will initially be up to 10 unscreened adult volunteers who have been previously studied on the 1.5-Tesla Signa scanner. Subjects will be required to provide informed consent, and to not have any medical exclusions as noted in the consent form and below, particularly metallic objects and/or pregnancy. Once procedures are optimized, up to 10 pediatric subjects will be studied. These pilot subjects will be derived from the normal control pool of subjects who have been previously studied on the 1.5-Tesla Signa scanner. Informed consent and signed assent will be required, with the same exclusions.

MONOZYGOTIC TWINS:

Subjects must be monozygotic twins (MZ) as confirmed by twin-similarity questionnaire and by molecular cheek swab testing by polymerase chain reaction short tandem repeat multiplex loci sets to find differences in the DNA types of the two co-twins. The primary test set includes nine to fourteen unlinked loci with a combined matching probability for siblings p less than .0001. Cases yielding a probability of twinship less than 0.99 are tested further to a total of 21 loci. Subjects may also be requested to participate in an associated genetic protocol (96-M-0060).

ADHD PROBANDS:

Monozygotic twin.

Aged 6 - 21 years.

DSM-IV diagnosis of ADHD (inattentive, hyperactive-impulsive and combined types).

Age adjusted dimensional ratings (Conners Rating Scales-Revised, or Strengths and Weaknesses of ADHD and Normal Behavior (SWAN)) hyperactivity/impulsivity greater than or equal to 95th percentile in affected twin.

Consent and assent obtained in writing.

NORMAL PEDIATRIC VOLUNTEERS:

Except for pilot subjects (up to 10 subjects), must be monozygotic twin.

Same age-range as probands.

Parent and teacher ratings within one SD of population means on ADHD/hyperactivity factors.

Consent and assent obtained in writing.

EXCLUSION CRITERIA:

ADHD PROBANDS:

Presence of other psychiatric disorders that can produce symptoms similar to ADHD (e.g., major depression, bipolar disorder, severe anxiety disorders, pervasive developmental disorders, psychotic disorders, post-traumatic stress disorder).

Presence of neuropsychiatric conditions that may confound evaluation of ADHD (e.g., Tourette's syndrome, obsessive-compulsive disorder, or PANDAS (pediatric autoimmune neuropsychiatric disorders associated with streptococcus).

Presence of metal objects, pregnancy, or inability to provide a specimen of urine or blood to rule out pregnancy in females over age 12.

Presence of alcohol and/or other substance abuse.

NORMAL PEDIATRIC VOLUNTEERS:

Presence of any psychiatric disorders on structured psychiatric interview (DICA-IV).

Presence of known genetic conditions.

Presence or history of medical conditions.

Presence of metal objects, pregnancy, or inability to provide a specimen to rule out pregnancy in females over age 12.

Presence of alcohol and/or other substance abuse.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120
Dates: Start 2001-01-12; Study Completion 2007-01-31

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Brandt KR, Hattery RR. MRI during pregnancy. Eur Radiol. 1997;7(6):821. doi: 10.1007/s003300050213. No abstract available. PMID 9228095